CLINICAL TRIAL: NCT03443765
Title: Serum 25(OH) Vitamin D and Total Serum Immunoglobulin E Levels in Patients With Pityriasis Alba
Status: Active, not recruiting | Type: Observational
Sponsor: Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan (Other Government)
Responsible Party: Principal Investigator, Svetlana Osipova, MD, PhD, DS, Professor, Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan
Other Study IDs: Project #002
Record Dates: First submitted 2018-02-16; First posted 2018-02-23 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Pityriasis Alba
MeSH Terms: conditions — Dandruff

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with Pityriasis alba
  Interventions: Diagnostic Test: Detection of Plasma levels of 25(OH) vitamin D by ELISA technique; Diagnostic Test: Detection of Total serum immunoglobulin E by ELISA technique
- Healthy participants (control group)
  Interventions: Diagnostic Test: Detection of Plasma levels of 25(OH) vitamin D by ELISA technique; Diagnostic Test: Detection of Total serum immunoglobulin E by ELISA technique

INTERVENTIONS:
Diagnostic Test: Detection of Plasma levels of 25(OH) vitamin D by ELISA technique — Five milliliters of peripheral venous blood sample will be taken (after 8-12 hours of fasting) from each participant and will be collected into HumaTube Serum Gel - C/A for ELISA. Serum will be appropriately obtained and stored at -20°C maximum of 30 days. Plasma levels of 25(OH) vitamin D will be detected by enzyme-linked immunosorbent assay (ELISA) technique.
Diagnostic Test: Detection of Total serum immunoglobulin E by ELISA technique — Five milliliters of peripheral venous blood sample will be taken (after 8-12 hours of fasting) from each participant and will be collected into HumaTube Serum Gel - C/A for ELISA. Serum will be appropriately obtained and stored at -20°C maximum of 30 days. Total serum immunoglobulin E will be detected by enzyme-linked immunosorbent assay (ELISA) technique.

SUMMARY:
Pityriasis alba (PA) is a common, benign skin disorder occurring predominantly in children and adolescents. It is characterized by ill-defined hypopigmented macules and patches, round or oval in shape. They are most commonly located on the face (especially the cheeks), arms, and upper trunk; and they are more noticeable in people with darker skin types. Sun exposure accentuates the lesions. Patients and their parents are often anxious about the cosmetic appearance of the lesions. PA is not seasonal, although peeling may be worse in the winter (as a result of dry air in homes) and lesions may be more obvious in the spring and summer (as a result of sun exposure and darkening of the surrounding skin).No specific cause of PA has been identified. It is not contagious, and no infectious etiology has been reported. It is most common in individuals with a history of atopy, although it may occur in nonatopic individuals.

In the present study, we will investigate the role of serum vitamin D levels and serum total IgE levels with development and course of PA. Plasma levels of 25(OH) vitamin D and Total serum immunoglobulin E will be determined by using ELISA technique.

DETAILED DESCRIPTION:
The prospective cohort study will be conducted on the basis of Research Institute of Epidemiology, Microbiology and Infectious Disease, Ministry of Public Health of the Republic of Uzbekistan.

Both informed and written consents will be obtained from the parents or from appropriate relative or guardian of the patients and healthy individuals of the control group.

Study participants will be included about 30 children aged 5 to 12 years with pityriasis alba. The control group will be included about 20 healthy individuals. All the participants will be residents of Uzbekistan.

Diagnosis of pityriasis alba Diagnosis of pityriasis alba will be based on the results of clinical examination. Inclusion criteria: revealing multiple round or oval-shaped hypopigmented macules or patches with indistinct margins. A weak erythema may be observed in some patches. The lesions number could varied from four to ten, 0.5 cm - 5 cm in size, and they are distributed predominantly on the face, neck, upper arms, and upper trunk.

Exclusion criteria The exclusion criteria: chronic and acute infectious diseases, endocrine diseases, congenital diseases, allergic dermatitis, bronchial asthma, allergic rhinitis and/or conjunctivitis, other skin disorders, history of using vitamin D supplements within three months ago, or use of any medication influencing endocrine parameters.

Measurement of anthropometric indices Demographic data will be obtained in the survey included age, gender, and body mass index (BMI) calculated as weight (kg)/height2 (m2).

Sample Collection and Storage Five milliliters of peripheral venous blood sample will be taken (after 8-12 hours of fasting) from each participant and will be collected into HumaTube Serum Gel - C/A for ELISA. Serum will be appropriately obtained and stored at -20°C maximum of 30 days. All blood samples will be collected during summer period.

Estimation of Vitamin D and Total Immunoglobulin E Plasma levels of 25(OH) vitamin D (DIAsource kit, Belgium) and Total serum immunoglobulin E (HUMAN kit, Germany) will be determined using ELISA technique.

Classification of Vitamin D and Total Immunoglobulin E Serum vitamin D level will be classified as reported by Holick (Holick MF. 2007). Levels of vitamin D ≤20, 21-29, ≥30-150, and >150 ng/ml will be considered as vitamin D deficiency, vitamin D insufficiency, vitamin D sufficiency and vitamin D intoxication, respectively.

Normal levels of total immunoglobulin E for children 1-6 years old - <30 Ul/ml, 7-9 years old - <60 Ul/ml and 10-12 years old - <100 Ul/ml, 13-16 years old - <150 Ul/ml.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Pityriasis alba
* Healthy individuals (control group)

Exclusion Criteria:

* chronic and acute infectious diseases;
* endocrine diseases;
* congenital diseases;
* allergic dermatitis;
* bronchial asthma;
* allergic rhinitis and/or conjunctivitis;
* other skin disorders;
* history of using vitamin D supplements within three months ago, or use of any medication influencing endocrine parameters.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The prospective cohort study will be conducted on the basis of Research Institute of Epidemiology, Microbiology and Infectious Disease, Ministry of Public Health of the Republic of Uzbekistan. All participants will be residents of Uzbekistan.
  Diagnosis of pityriasis alba will be based on the results of clinical examination.
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum 25(OH) vitamin D levels in the patients with pityriasis alba | up to 24 months
  In this study we expect to determine a role of Vitamin D in the development and course of pityriasis alba
Total serum immunoglobulin E levels in the patients with pityriasis alba | up to 24 months
  In this study we expect to determine a role of immunoglobulin E in the development and course of pityriasis alba

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Osipova, MD, PhD, DS, Principal Investigator — research institute of epidemiology, microbiology and infectious diseases
Locations (1):
- Research institute of epidemiology, microbiology and infectious diseases, Tashkent, Uchtepa, Uzbekistan

REFERENCES:
- [Background] Toychiev A, Mirzoeva M, Davis N, Islamova J, Osipova S. Pityriasis alba: Possible associations with intestinal helminths and pathogenic protozoa. Int J Clin Pract. 2020 Feb;74(2):e13441. doi: 10.1111/ijcp.13441. Epub 2019 Oct 30. PMID 31633268